CLINICAL TRIAL: NCT00260000
Title: Study of the Response of Tetrahydrobiopterin on S-Phenylalanine in Patients With PKU Housing the Y414C Mutation
Brief Title: Study of BH4, a New and Simple Treatment of Mild PKU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Kennedy Institute-National Eye Clinic (Other Government)
Collaborators: Sygekassernes Helsefond (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2612-2706-BH4-1
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2006-04-13 (Estimated); Status verified 2006-04

CONDITIONS: Phenylketonuria
Keywords: mild PKU; Y414C; 5,6,7,8-tetrahydrobiopterin, BH4; treatment without protein restriction
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

INTERVENTIONS:
Drug: 5,6,7,8-tetrahydrobiopterin

SUMMARY:
The main purpose is to test whether treatment with BH4-tablets can replace the protein restrictive diet in patients with mild PKU caused by a certain frequent mutation.

DETAILED DESCRIPTION:
PKU, phenylketonuria, is a rare, inherited metabolic disorder that results in mental retardation if not a very strict low-protein diet is started within the first weeks of life.

The conversion of phenylalanine, phe, to tyrosine is defect, phe accumulates, leading to brain damage. There are different degrees of severity, reflecting the spectrum of mutant genes. BH4, tetrahydrobiopterin, is a co-enzym for the conversion of phe to tyrosine. It is known that BH4 can lower phe in some patients with milder forms of PKU.

The main purpose is to test whether treatment with oral BH4 can replace the protein restrictive diet in patients with mild PKU caused by the frequent mutation Y414C in the phenylalanine hydroxylase gene.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed mild PKU with 2 known mutations in the PAH gene, hereof at least one Y414C From the age of eight Informed consent -

Exclusion Criteria:

Less than 8 years of age Pregnancy or treated with the intensive diet of pregnancy

-

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 2005-04; Study Completion 2005-12

PRIMARY OUTCOMES:
Fasting S-phenylalanine at day 0, 1, 2, 5, 7 in each week of treatment with BH4.

CONTACTS AND LOCATIONS:
Overall Officials: Jytte B Nielsen, DMSc, Principal Investigator — The Kennedy Institute-National Eye Clinic
Locations (1):
- The Kennedy Institute-National Eye Clinic, Glostrup Municipality, Copenhagen, Denmark